CLINICAL TRIAL: NCT04782297
Title: Post-Market Clinical Follow-up Study - Open Label, Consecutive Series, Observational Study on the Use of Medcomp Long Term Catheters for Hemodialysis (LTHD)
Brief Title: Long Term Hemodialysis Catheters (LTHD) Post Market Clinical Follow up (PMCF)
Acronym: LTHD PMCF
Status: Withdrawn | Type: Observational
Why Stopped: Recruitment and enrollment was not prioritized by sites and no enrollments occurred over the course of 1 year.
Sponsor: Medical Components, Inc dba MedComp (Industry)
Collaborators: Syneos Health (Other); Veeva Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: PMCF_LTHD_201
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: CKD; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Titan HD Catheter: The Titan HD Catheter is a double lumen catheter that provides 2 dedicated (arterial/venous) access lumens. Each lumen is connected through an extension line with female luer connectors. The arterial and venous catheter lumens connect to a hub to facilitate connection of extension tubes with clamps intended to prevent air/fluid communication and control fluid flow through the catheter. At the proximal end of the extension tubes are female Luer fittings to provide a needleless connection. The clamps and the sleeves are color-coded red for the arterial lumen and blue for the venous lumen. Each catheter has a cuff which is intended to be positioned underneath the skin at the skin exit to aid in securing the catheter and to provide a barrier to minimize the risk of infection. Each lumen is connected through an extension line with female Luer connectors. The transition between lumen and extension is housed within a molded hub.
  Interventions: Device: Long term hemodialysis catheter
- Hemo-Flow Catheter: The Hemo-Flow® Catheter has two lumens (one arterial lumen, one venous lumen) comprised of a biocompatible polymeric material that contains radiopaque filler to allow radiographic imaging of the distal tips to ensure proper placement into the superior vena cava. The arterial lumen is utilized to withdraw blood from the patient and the venous lumen returns the blood to the patient after treatment
  Interventions: Device: Long term hemodialysis catheter

INTERVENTIONS:
Device: Long term hemodialysis catheter — There will be no interventions in this study. Strictly observational.

SUMMARY:
The primary objective of this observational PMCF study is to collect clinical data on the safety and efficacy of Medcomp Long Term Hemodialysis (LTHD) Catheter Kits in compliance with MDR 2017/745.

DETAILED DESCRIPTION:
The Observational Study will enroll a target of 198 subjects across two cohorts of 89 patients per cohort, with each cohort representing one catheter type. Retrospective patients previously treated with either a Hemo-Flow or Titan HD catheter will be enrolled. The primary endpoint of this study for all device families is insertion success. For the purposes of this data, a successful insertion will be defined as the successful initiation of vascular access device insertion, as determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of enrollment
2. Patients who have previously received the Medcomp subject device or patients currently receiving hemodialysis treatment, who have had a Medcomp subject device implanted for >90 days
3. Health records relevant to this study are complete and accessible by Study team at the hemodialysis center, implantation center, medical facilities where complications are treated, and by the participating Principal Investigator (PI)
4. Subject or authorized representative participated in the Informed Consent process and signed/dated the relevant institutional ethics committee approved Informed Consent form

Exclusion Criteria:

1. Meet any of the contraindications listed on the Medcomp Long Term Hemodialysis Catheter Instructions for Use
2. Participation in any other drug, device, or biologic study concomitantly, or within the last 30 days (which may clinically interfere with this Study in the opinion of the sponsor in consultation with the Principal Investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective patients (those who already have one of the Medcomp LTHD catheters inserted) will be enrolled. Retrospective patients from the previous 36 months will be approached for participation in the study. Patients who have previously received a Medcomp LTHD catheter will also be approached for consent and assessment of eligibility.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-30 (Estimated); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Insertion Success | Percentage at Insertion
  Successful initiation of vascular access device insertion, as determined by the investigator.

SECONDARY OUTCOMES:
Adverse Events (Infection per 1000 catheter days) | 1000 catheter days
  Infection, Removals due to infection or thrombosis, catheter related blood stream infection (CRBSI)

CONTACTS AND LOCATIONS:
Locations (2):
- University of Maryland School of Medicine Vascular & Interventional Radiology Department, Baltimore, Maryland, United States
- Hospital Universitari Arnau de Vilanova, Lleida, Spain